CLINICAL TRIAL: NCT07191379
Title: Self-administered Subcutaneous Daratumumab in Patients With Multiple Myeloma. An Open Label, Phase Four, Prospective, Non-randomized, Sponsor-initiated Multicenter Feasibility Study
Brief Title: Self-administered Subcutaneous Daratumumab in Patients With Multiple Myeloma
Acronym: SCILLA
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Odense University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SCILLA
Record Dates: First submitted 2025-09-09; First posted 2025-09-24 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Multiple Myeloma in Relapse
Keywords: Treatment at home; Daratumumab; Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Intervention Model Description: It is a feasibility study assessing the feasibility and safety of self-administration of SC daratumumab in the homes of the patients. The study intervention is self-administration of SC daratumumab by the patient, thereby changing the administration from an outpatient setting to a home setting. To reduce potential bias, patients will function as their own controls by receiving alternating treatments at home and in the outpatient clinic. To participate, patients must be scheduled for SC daratumumab alone or in combination with other drugs not necessitating outpatient visits on days of planned SC daratumumab self-administration
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Self-administration of SC daratumumab by the patient at their own home (Experimental): The study intervention is self-administration of SC daratumumab by the patient, thereby changing the administration from an outpatient setting to a home setting. To reduce potential bias, patients will function as their own controls by receiving alternating treatments at home and in the outpatient clinic.
  Interventions: Other: The study intervention is self-administration of SC daratumumab by the patient, thereby changing the administration from an outpatient setting to a home setting.

INTERVENTIONS:
Other: The study intervention is self-administration of SC daratumumab by the patient, thereby changing the administration from an outpatient setting to a home setting. — The study intervention is self-administration of SC daratumumab by the patient, thereby changing the administration from an outpatient setting to a home setting. To reduce potential bias, patients will function as their own controls by receiving alternating treatments at home and in the outpatient clinic.

SUMMARY:
The main goal in this open label, phase four, prospective, non-randomized, sponsor-initiated multicenter feasibility study is to evaluate the feasibility and safety of self-administration of subcutaneously (SC) daratumumab in the patients with multiple myeloma in their own home. The study intervention is self-administration of SC daratumumab by the patient, thereby changing the administration from an outpatient setting to a home setting. To reduce potential bias, patients will function as their own controls by receiving alternating treatments at home and in the outpatient clinic. To participate, patients must be scheduled for SC daratumumab alone or in combination with other drugs not necessitating outpatient visits on days of planned SC daratumumab self-administration. Patients can be included and trained during cycle 1 and 2, but only treatments administered in cycle 3-6 are considered protocol treatments. Here, patients will receive SC daratumumab once every second week with treatments at day 1 administered in the outpatient clinic and treatments at day 15 administered at home. From cycle 7 onwards, patients continues SC daratumumab outside protocol according to local standards.

At inclusion, baseline demographic and clinical data should be registered for included patients. For each SC daratumumab administration in the protocol, planned treatment location (home/hospital) should be registered together with information on whether the dose was administered as planned. For each protocol treatment, regardless of treatment location, patients, caregivers, and healthcare professionals should register their time spent. In addition, patients should complete the Health Literacy Questionnaire (HLQ) and caregivers are to complete the Caregiver Roles and Responsibilities Scale (CRRS). Throughout the study, patient will also register all unplanned contacts to the healthcare system. Patient will also be asked to complete an evaluation form. Lastly, qualitative evaluations of the experience of self-administration will be conducted through semi-structured interviews with patients and caregivers, as well as focus group interviews with involved healthcare professionals.

DETAILED DESCRIPTION:
Introduction Subcutaneous (SC) daratumumab has significantly improved outcomes for patients with multiple myeloma (MM), allowing for longer survival with continuous treatment. However, this has also increased the burden on outpatient clinics. Future demographic shifts-more elderly and fewer healthcare workers-will only worsen the situation. For patients, ongoing treatment often means long, tiring trips to the hospital and increased infection risks. Home treatment may solve these issues.

Previous studies have shown that SC daratumumab administered at home by healthcare staff is safe and convenient, and that patients-even elderly ones-can successfully self-administer SC medications like bortezomib. In Denmark, some hospitals already offer self-administration of SC daratumumab, but without systematic data collection.

This study aims to evaluate the feasibility, safety, efficiency, and cost-effectiveness of home-based, self-administered SC daratumumab within a structured, prospective framework.

Background

Target Population:

MM is the second most common hematologic cancer, with ~350 new cases annually in Denmark. The median age at diagnosis is 69, and ~30% are of working age. Survival has doubled over the past 20 years, but the disease remains incurable and requires lifelong treatment.

Daratumumab Treatment:

Daratumumab, a key anti-CD38 antibody in MM treatment, was originally IV but is now available as SC, enabling administration outside the hospital.

Home-Based Treatment:

Home administration reduces infection risk and travel burden-particularly important during the COVID-19 era. Studies show improved quality of life (QoL) and reduced healthcare costs (up to 50%) with self-administration. Given workforce shortages in healthcare, shifting eligible treatments to the home may help relieve system pressure.

Risk and Benefit Assessment SC daratumumab is well-established, with a known safety profile. The only change in this study is shifting administration from healthcare professionals to patients. Potential risks (e.g. incorrect administration) are mitigated through a structured training program, written instructions, and continuous support. Benefits include greater autonomy, fewer hospital visits, and resource savings. The study is considered low-risk and ethically justified.

Study Population 50 MM patients scheduled for SC daratumumab treatment and considered eligible for self-administration.

Interview Sampling:

15 patients with caregivers and 2-3 healthcare professionals per site.

Study Design and Procedures A phase IV, multicenter, prospective, non-randomized feasibility study using mixed methods. Patients will alternate between outpatient (day 1) and home (day 15) treatment during cycles 3-6.

Patients will be trained by nurses using standardized materials until they and the nurse agree the patient is confident in self-administration.

Study Treatment SC daratumumab will be administered according to national guidelines. During cycles 3-6, patients will receive treatment on day 1 in clinic and self-administer at home on day 15. Medication and instructions will be provided at the clinic. Before each home administration, a nurse will confirm eligibility via phone.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with MM
* Initiating treatment with SC daratumumab
* Able to read and understand the Danish language
* Are considered suitable for self-administration of SC daratumumab at home (in the opinion of the healthcare professional)
* Willing and able to complete questionnaires and participate in an interview

Exclusion Criteria:

* Resident on an unbridged island
* Receiving co-treatment with other anti-myeloma treatments necessitating hospitals visits on days of home administration
* Anything related to their ability to self-administer SC daratumumab at home e.g. physical inabilities or cognitive impairment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
To evaluate the feasibility of self-administration of SC daratumumab in the patients´ homes | 12 months
  * Number of doses given unplanned/outside indication
  * Number of doses administered as planned at home and at the hospital

SECONDARY OUTCOMES:
To evaluate the feasibility of self-administration of SC daratumumab in the patients´ homes | 12 months
  - Number of discarded doses
To evaluate the safety of self-administration of SC daratumumab in the patients' home | 12 month
  - numbers of unexpected serious adverse events
To evaluate the feasibility of self-administration of SC daratumumab in the patients´ homes | 12 months
  * Number of patients willing to participate, dropping out, and/or deemed ineligible to participate
  * Reasons for this
To evaluate costs related to self-administration of SC daratumumab in the patients' home compared to traditional administration at the outpatient clinic | 12 months
  - Time spent by patients, caregivers, and healthcare professionals administering the treatment in minutes
To evaluate patients' satisfaction with self-administration of SC daratumumab | 12 months
  Satisfaction scores collected via patient-reported outcomes (PRO)
Perspectives on treatment at home of patients, caregivers, and healthcare staff | 14 months
  Semi-structured joint interviews with patients and their caregivers after completing the four treatment cycles under protocol defined conditions and a focus group interviews with involved healthcare professionals at end of study.
To evaluate the feasibility of self-administration of SC daratumumab in the patients´ homes | 12 months
  - Reasons for discarding doses

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Lund, MD, Principal Investigator — Vejle Hospital

IPD SHARING:
Plan to Share IPD: No
Not mandatory.